CLINICAL TRIAL: NCT06255327
Title: The Effectiveness of The "I Cough" Care Program to Dyspnea, Respiratory Parameters, Mobility and Pain After Major Abdominal Surgery.
Brief Title: Effectiveness of I COUGH Program to Dyspnea, Respiratory Parameters, Mobility and Pain After Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: YTU.PT.TH.01/2023
Record Dates: First submitted 2023-12-25; First posted 2024-02-13 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Dyspnea; Pain; Respiratory Insufficiency; Mobility Limitation
Keywords: I COUGH; Dyspnea; Respiratory Parameters; Pain; Major Abdominal Surgery
MeSH Terms: conditions — Dyspnea; Pain; Respiratory Insufficiency; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: The sample of the study (n=60) consisted of patients underwent major abdominal surgery required general anesthesia and hospital stay who got diagnosed by consultant general and bariatric surgery, being between 30-60 years old (39.9±8.82 years old; 47 F/ 13 M) volunteered to attend this study. The participants were randomly divided into two groups.
Who Masked: Participant
Masking Description: Participants in the control group were not given any information or training before or after the operation, and they were on routine hospital care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group participants underwent evaluations on the first day after 10 hours following surgery and, on the day, they were discharged from the clinic, by using pulse oximetry, sphygmometer, spirometry tests, VAS, MBDS and activity and mobility promotion (AMP). Participants in the control group were not given any information or training before or after the operation, and they were on routine hospital care.
- Experimental group (Experimental): The participants in the experimental group underwent the application of I COUGH (Incentive spirometry, Coughing/Deep breathing, Oral care, Understanding (Education of patient and family), Getting out of bed, and raising the Head of the bed). The participants underwent evaluations on the first day after 10 hours following surgery and, on the day, they were discharged from the clinic. Including Pulse Oximetry, Sphygmometer, Spirometry Tests, VAS, MBDS, AMP.
  Interventions: Other: I COUGH care program

INTERVENTIONS:
Other: I COUGH care program — The I COUGH program, initiated 10 hours after surgery, emphasizes the following elements:
  Incentive spirometry: Encouraging patients to use the Flow-IS device ten times every two hours for three days.
  Coughing and deep breathing: Participants should perform 3-5 coughs and deep breaths every 2 hours for 3 days.
  Oral care: Brushing teeth and using mouthwash twice daily between 8:00 a.m. and 8:00 p.m. Mouth brushes should be sterile, and non-alcoholic mouthwash is recommended.
  Understanding (education): Patients and their relatives receive instructions on the care program and steps to follow.
  Getting out of bed: Patients are encouraged to sit in a chair at least once and walk at least 3 times per day in the room and corridor with assistance as needed.
  Head-of-bed elevation: Keeping the head of the bed elevated more than 30 degrees.
  Arms: Experimental group

SUMMARY:
The purpose of the current study was to investigate the effect of the I COUGH care program following major abdominal surgery dyspnea, oxygen saturation, pulmonary function, mobility, and pain after major abdominal surgery (MAS), participants were subjected to the "I COUGH" care program designed to support their health condition and reduce complications. The study aimed to investigate a simple and inexpensive pulmonary care program that can be easily understood and remembered by patients, their families, and medical staff.

Ho: The I COUGH care program after MAS does not improves pulmonary functions, oxygen saturation, mobility and decrease dyspnea and pain after MAS.

H1: The I COUGH care program improves pulmonary functions, oxygen saturation mobility and decrease dyspnea and pain after MAS.

DETAILED DESCRIPTION:
A total of 60 adult individuals aged between 30 and 60 years (mean age of 39.9±8.82) comprising 13 males and 47 females underwent major abdominal surgery requiring general anesthesia and hospitalization were invited to study. Patients were randomly assigned to either the Control Group (CG, n=30) or the Experimental Group (EG, n=30) using the block randomization method. Patients in the EG participated in the I COUGH care program included flow-incentive spirometer, oral care, coughing and breathing exercises, patient, and family education, getting out of bed, and elevating the head of the bed by more than 30 degrees for 3 days post-surgery. The patients in the CG did not undergo any interventions. All participants were assessed in terms of vital signs as heart rate, blood pressure, respiratory rate, and oxygen saturation. Moreover, dyspnea was assessed using the Modified Borg dyspnea Scale, pulmonary functions were evaluated using spirometry, mobility was assessed by Activity and Mobility Promotion scale and pain assessed Visual Analog Scale. Data were collected from all patients at baseline 10 h after the first day of surgery and on the day of discharge from the hospitals. The findings of the present study revealed that the I COUGH care program effectively improved pulmonary function and blood oxygenation, reduced the incidence of dyspnea, increased mobility, and decreased postoperative pain, with a statistically significant difference between the experimental and control groups (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Eligible patients are adults of both sexes between 30-60 years (Through the study, we are trying to reduce the variance and confounding factors that may arise from including patients who are less than 30 years old due to different stages of growth, physical abilities, hormonal levels, etc., or over 60 years old due to the prevalence of chronic diseases or diseases associated with aging).
* Patients underwent elective abdominal surgery that required general anaesthesia and hospital stay e.g., Hernia repair, gall bladder removal, exploratory laparotomy, morbid obesity, ovarian cyst, Sigmoid diverticulitis, appendicitis, or other abdominal cavity procedures performed by laparoscopy and conventional laparotomy with a 5 cm or less incision above or extending above the umbilicus. (Incisions > 5cm may affect on possible results might be impacted in terms of: Increased risk of infection, risk of bleeding, pain, and discomfort during ambulation).

Exclusion Criteria:

* The patient complains of an unstable heart rate or cardiac condition.
* Symptomatic heart failure, unstable angina.
* Pulmonary Hypertension
* Unstable hypertension
* The patient underwent organ transplants.
* The patient presented an aneurysm of any arterial segment.
* Serious condition or transferred to the intensive care unit after surgery.
* Severe nephropathy.
* A patient with cancer.
* Cerebrovascular accident / Stroke.
* Patient with balance or vestibular disorder.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate (HR) | 3 days of postoperatively
  The number of heart beats per minute.
Systolic Blood pressure (SBP) | 3 days of postoperatively
  The minimum pressure recorded just prior to the next contraction.
Diastolic Blood pressure (DBP) | 3 days of postoperatively
  The maximum blood pressure during contraction of the ventricles.
Respiratory Rate (RR) | 3 days of postoperatively
  The number of breaths they take per minute.
Oxygen Saturation (SPO2) | 3 days of postoperatively
  A pulse oximeter reading that indicates what percentage of your blood is saturated.
Modified Borg Dyspnea Scale (MBDS) | 3 days of postoperatively
  A valid and reliable tool to measure the intensity of dyspnea. It is a categorical scale with ratio properties, rating from 0 to 10, 0 being not dyspneic at all and 10 being maximally dyspneic.
Pulmonary Function Test FVC | 3 days of postoperatively
  Noninvasive test that show how well the lungs are working, measuring of FVC
Pulmonary Function Test FEV | 3 days of postoperatively
  Noninvasive tests that show how well the lungs are working, measuring of FEV
Pulmonary Function Test FEV1/FVC | 3 days of postoperatively
  Noninvasive tests that show how well the lungs are working, measuring of FEV1/FVC
Pulmonary Function Test PEFR | 3 days of postoperatively
  Noninvasive tests that show how well the lungs are working, measuring of PEFR.
Activity and Mobility Promotion (AMP) | 3 days of postoperatively
  AMP is based on measuring increasing patient mobility during hospital stay. The initial goals of this program included mobilization of each patient 3 times per day, documentation of patient mobility levels on the AMP scale.
Visual Analogue Scale (VAS) | 3 days of postoperatively
  This measure is based on self-reported symptoms and is recorded with a single mark placed along a 10-cm line, which represents a continuum between "no pain" on the left end (0 cm) and "worst pain" on the right end. to determine the intensity of pain and its enhancement when coughing in the postoperative area.

CONTACTS AND LOCATIONS:
Overall Officials: Feras M Tana, MSc, Principal Investigator — Yeditepe University
Locations (3):
- Libya (3):
  - AL-ASSEMA Hospital, Tripoli
  - AL-KHALIL Hospital, Tripoli
  - ROYAL Clinic, Tripoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branson RD. The scientific basis for postoperative respiratory care. Respir Care. 2013 Nov;58(11):1974-84. doi: 10.4187/respcare.02832. PMID 24155356
- [Background] Moore JA, Conway DH, Thomas N, Cummings D, Atkinson D. Impact of a peri-operative quality improvement programme on postoperative pulmonary complications. Anaesthesia. 2017 Mar;72(3):317-327. doi: 10.1111/anae.13763. Epub 2017 Jan 4. PMID 28054356
- [Background] Smetana GW. Postoperative pulmonary complications: an update on risk assessment and reduction. Cleve Clin J Med. 2009 Nov;76 Suppl 4:S60-5. doi: 10.3949/ccjm.76.s4.10. PMID 19880838
- [Background] Odor PM, Bampoe S, Gilhooly D, Creagh-Brown B, Moonesinghe SR. Perioperative interventions for prevention of postoperative pulmonary complications: systematic review and meta-analysis. BMJ. 2020 Mar 11;368:m540. doi: 10.1136/bmj.m540. PMID 32161042
- [Background] Boden I, Skinner EH, Browning L, Reeve J, Anderson L, Hill C, Robertson IK, Story D, Denehy L. Preoperative physiotherapy for the prevention of respiratory complications after upper abdominal surgery: pragmatic, double blinded, multicentre randomised controlled trial. BMJ. 2018 Jan 24;360:j5916. doi: 10.1136/bmj.j5916. PMID 29367198
- [Background] Brooks-Brunn JA. Predictors of postoperative pulmonary complications following abdominal surgery. Chest. 1997 Mar;111(3):564-71. doi: 10.1378/chest.111.3.564. PMID 9118688
- [Background] Manzano RM, Carvalho CR, Saraiva-Romanholo BM, Vieira JE. Chest physiotherapy during immediate postoperative period among patients undergoing upper abdominal surgery: randomized clinical trial. Sao Paulo Med J. 2008 Sep;126(5):269-73. doi: 10.1590/s1516-31802008000500005. PMID 19099160
- [Background] Fagevik Olsen M, Hahn I, Nordgren S, Lonroth H, Lundholm K. Randomized controlled trial of prophylactic chest physiotherapy in major abdominal surgery. Br J Surg. 1997 Nov;84(11):1535-8. doi: 10.1111/j.1365-2168.1997.02828.x. PMID 9393272
- [Background] Siafakas NM, Mitrouska I, Bouros D, Georgopoulos D. Surgery and the respiratory muscles. Thorax. 1999 May;54(5):458-65. doi: 10.1136/thx.54.5.458. No abstract available. PMID 10212115
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Cheifetz O, Lucy SD, Overend TJ, Crowe J. The effect of abdominal support on functional outcomes in patients following major abdominal surgery: a randomized controlled trial. Physiother Can. 2010 Summer;62(3):242-53. doi: 10.3138/physio.62.3.242. Epub 2010 Jul 23. PMID 21629603
- [Background] Smith PR, Baig MA, Brito V, Bader F, Bergman MI, Alfonso A. Postoperative pulmonary complications after laparotomy. Respiration. 2010;80(4):269-74. doi: 10.1159/000253881. Epub 2009 Oct 28. PMID 19864881
- [Background] Lawrence VA, Hilsenbeck SG, Mulrow CD, Dhanda R, Sapp J, Page CP. Incidence and hospital stay for cardiac and pulmonary complications after abdominal surgery. J Gen Intern Med. 1995 Dec;10(12):671-8. doi: 10.1007/BF02602761. PMID 8770719
- [Background] Nafiu OO, Ramachandran SK, Ackwerh R, Tremper KK, Campbell DA Jr, Stanley JC. Factors associated with and consequences of unplanned post-operative intubation in elderly vascular and general surgery patients. Eur J Anaesthesiol. 2011 Mar;28(3):220-4. doi: 10.1097/EJA.0b013e328342659c. PMID 21191304
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Sabate S, Mazo V, Canet J. Predicting postoperative pulmonary complications: implications for outcomes and costs. Curr Opin Anaesthesiol. 2014 Apr;27(2):201-9. doi: 10.1097/ACO.0000000000000045. PMID 24419159
- [Background] Davies SJ, Francis J, Dilley J, Wilson RJ, Howell SJ, Allgar V. Measuring outcomes after major abdominal surgery during hospitalization: reliability and validity of the Postoperative Morbidity Survey. Perioper Med (Lond). 2013 Feb 4;2(1):1. doi: 10.1186/2047-0525-2-1. PMID 24472150
- [Background] So MW, Heo HM, Koo BS, Kim YG, Lee CK, Yoo B. Efficacy of incentive spirometer exercise on pulmonary functions of patients with ankylosing spondylitis stabilized by tumor necrosis factor inhibitor therapy. J Rheumatol. 2012 Sep;39(9):1854-8. doi: 10.3899/jrheum.120137. Epub 2012 Aug 1. PMID 22859343
- [Background] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401
- [Background] Tyson AF, Kendig CE, Mabedi C, Cairns BA, Charles AG. The effect of incentive spirometry on postoperative pulmonary function following laparotomy: a randomized clinical trial. JAMA Surg. 2015 Mar 1;150(3):229-36. doi: 10.1001/jamasurg.2014.1846. PMID 25607594
- [Background] Nishikawa M, Honda M, Kimura R, Kobayashi A, Yamaguchi Y, Hori S, Kobayashi H, Waragai M, Kawamura H, Nakayama Y, Todate Y, Takano Y, Yamaguchi H, Hamada K, Iketani S, Seto I, Izumi Y, Seto K. The bacterial association with oral cavity and intra-abdominal abscess after gastrectomy. PLoS One. 2020 Nov 9;15(11):e0242091. doi: 10.1371/journal.pone.0242091. eCollection 2020. PMID 33166362
- [Background] Cassidy MR, Rosenkranz P, McCabe K, Rosen JE, McAneny D. I COUGH: reducing postoperative pulmonary complications with a multidisciplinary patient care program. JAMA Surg. 2013 Aug;148(8):740-5. doi: 10.1001/jamasurg.2013.358. PMID 23740240
- [Background] Tazreean R, Nelson G, Twomey R. Early mobilization in enhanced recovery after surgery pathways: current evidence and recent advancements. J Comp Eff Res. 2022 Feb;11(2):121-129. doi: 10.2217/cer-2021-0258. Epub 2022 Jan 20. PMID 35045757
- [Background] Cassidy MR, Rosenkranz P, Macht RD, Talutis S, McAneny D. The I COUGH Multidisciplinary Perioperative Pulmonary Care Program: One Decade of Experience. Jt Comm J Qual Patient Saf. 2020 May;46(5):241-249. doi: 10.1016/j.jcjq.2020.01.005. Epub 2020 Jan 30. PMID 32122711
- [Background] Weindler J, Kiefer RT. The efficacy of postoperative incentive spirometry is influenced by the device-specific imposed work of breathing. Chest. 2001 Jun;119(6):1858-64. doi: 10.1378/chest.119.6.1858. PMID 11399715
- [Background] Banerjee D, Kamuren J, Baird GL, Palmisciano A, Krishnan I, Whittenhall M, Klinger JR, Ventetuolo CE. The Modified Borg Dyspnea Scale does not predict hospitalization in pulmonary arterial hypertension. Pulm Circ. 2017 Apr-Jun;7(2):384-390. doi: 10.1177/2045893217695568. Epub 2017 Mar 16. PMID 28597751
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] McLaughlin KH, Friedman M, Hoyer EH, Kudchadkar S, Flanagan E, Klein L, Daley K, Lavezza A, Schechter N, Young D; JH-AMP Group. The Johns Hopkins Activity and Mobility Promotion Program: A Framework to Increase Activity and Mobility Among Hospitalized Patients. J Nurs Care Qual. 2023 Apr-Jun 01;38(2):164-170. doi: 10.1097/NCQ.0000000000000678. Epub 2022 Dec 3. PMID 36729980
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Hedenstierna G, Rothen HU. Respiratory function during anesthesia: effects on gas exchange. Compr Physiol. 2012 Jan;2(1):69-96. doi: 10.1002/cphy.c080111. PMID 23728971
- [Background] Hall JC, Tarala RA, Tapper J, Hall JL. Prevention of respiratory complications after abdominal surgery: a randomised clinical trial. BMJ. 1996 Jan 20;312(7024):148-52; discussion 152-3. doi: 10.1136/bmj.312.7024.148. PMID 8563533
- [Background] Wren SM, Martin M, Yoon JK, Bech F. Postoperative pneumonia-prevention program for the inpatient surgical ward. J Am Coll Surg. 2010 Apr;210(4):491-5. doi: 10.1016/j.jamcollsurg.2010.01.009. PMID 20347742
- [Background] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Background] Lawrence VA, Cornell JE, Smetana GW; American College of Physicians. Strategies to reduce postoperative pulmonary complications after noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):596-608. doi: 10.7326/0003-4819-144-8-200604180-00011. PMID 16618957
- [Background] Pasquina P, Tramer MR, Granier JM, Walder B. Respiratory physiotherapy to prevent pulmonary complications after abdominal surgery: a systematic review. Chest. 2006 Dec;130(6):1887-99. doi: 10.1378/chest.130.6.1887. PMID 17167013
- [Background] Weller WE, Rosati C. Comparing outcomes of laparoscopic versus open bariatric surgery. Ann Surg. 2008 Jul;248(1):10-5. doi: 10.1097/SLA.0b013e31816d953a. PMID 18580201
- [Background] Sum SK, Peng YC, Yin SY, Huang PF, Wang YC, Chen TP, Tung HH, Yeh CH. Using an incentive spirometer reduces pulmonary complications in patients with traumatic rib fractures: a randomized controlled trial. Trials. 2019 Dec 30;20(1):797. doi: 10.1186/s13063-019-3943-x. PMID 31888765
- [Background] Louie A, Feiner JR, Bickler PE, Rhodes L, Bernstein M, Lucero J. Four Types of Pulse Oximeters Accurately Detect Hypoxia during Low Perfusion and Motion. Anesthesiology. 2018 Mar;128(3):520-530. doi: 10.1097/ALN.0000000000002002. PMID 29200008
- [Background] Crisafulli E, Clini EM. Measures of dyspnea in pulmonary rehabilitation. Multidiscip Respir Med. 2010 Jun 30;5(3):202-10. doi: 10.1186/2049-6958-5-3-202. PMID 22958431
- [Background] Katz S, Arish N, Rokach A, Zaltzman Y, Marcus EL. The effect of body position on pulmonary function: a systematic review. BMC Pulm Med. 2018 Oct 11;18(1):159. doi: 10.1186/s12890-018-0723-4. PMID 30305051
- [Background] Spahija J, Marchie Md, Ghezzo H, Grassino A. Factors discriminating spontaneous pursed-lips breathing use in patients with COPD. COPD. 2010 Aug;7(4):254-61. doi: 10.3109/15412555.2010.496820. PMID 20673034
- [Background] Delgado HR, Braun SR, Skatrud JB, Reddan WG, Pegelow DF. Chest wall and abdominal motion during exercise in patients with chronic obstructive pulmonary disease. Am Rev Respir Dis. 1982 Aug;126(2):200-5. doi: 10.1164/arrd.1982.126.2.200. PMID 7103243
- [Background] Sharp JT, Drutz WS, Moisan T, Foster J, Machnach W. Postural relief of dyspnea in severe chronic obstructive pulmonary disease. Am Rev Respir Dis. 1980 Aug;122(2):201-11. doi: 10.1164/arrd.1980.122.2.201. No abstract available. PMID 7416599
- [Background] O'Neill S, McCarthy DS. Postural relief of dyspnoea in severe chronic airflow limitation: relationship to respiratory muscle strength. Thorax. 1983 Aug;38(8):595-600. doi: 10.1136/thx.38.8.595. PMID 6612651
- [Background] Kumar AS, Alaparthi GK, Augustine AJ, Pazhyaottayil ZC, Ramakrishna A, Krishnakumar SK. Comparison of Flow and Volume Incentive Spirometry on Pulmonary Function and Exercise Tolerance in Open Abdominal Surgery: A Randomized Clinical Trial. J Clin Diagn Res. 2016 Jan;10(1):KC01-6. doi: 10.7860/JCDR/2016/16164.7064. Epub 2016 Jan 1. PMID 26894090
- [Background] Grams ST, Ono LM, Noronha MA, Schivinski CI, Paulin E. Breathing exercises in upper abdominal surgery: a systematic review and meta-analysis. Rev Bras Fisioter. 2012 Sep-Oct;16(5):345-53. doi: 10.1590/s1413-35552012005000052. Epub 2012 Oct 9. PMID 23060237
- [Background] Thomas JA, McIntosh JM. Are incentive spirometry, intermittent positive pressure breathing, and deep breathing exercises effective in the prevention of postoperative pulmonary complications after upper abdominal surgery? A systematic overview and meta-analysis. Phys Ther. 1994 Jan;74(1):3-10; discussion 10-6. doi: 10.1093/ptj/74.1.3. PMID 8265725
- [Background] Sullivan KA, Churchill IF, Hylton DA, Hanna WC. Use of Incentive Spirometry in Adults following Cardiac, Thoracic, and Upper Abdominal Surgery to Prevent Post-Operative Pulmonary Complications: A Systematic Review and Meta-Analysis. Respiration. 2021;100(11):1114-1127. doi: 10.1159/000517012. Epub 2021 Jul 16. PMID 34274935
- [Background] Rowley DD, Malinowski TP, Di Peppe JL, Sharkey RM, Gochenour DU, Enfield KB. A Randomized Controlled Trial Comparing Two Lung Expansion Therapies After Upper Abdominal Surgery. Respir Care. 2019 Oct;64(10):1181-1192. doi: 10.4187/respcare.06812. Epub 2019 May 21. PMID 31113857
- [Background] Westwood K, Griffin M, Roberts K, Williams M, Yoong K, Digger T. Incentive spirometry decreases respiratory complications following major abdominal surgery. Surgeon. 2007 Dec;5(6):339-42. doi: 10.1016/s1479-666x(07)80086-2. PMID 18080608
- [Background] Spadaro S, Caramori G, Rizzuto C, Mojoli F, Zani G, Ragazzi R, Valpiani G, Dalla Corte F, Marangoni E, Volta CA. Expiratory Flow Limitation as a Risk Factor for Pulmonary Complications After Major Abdominal Surgery. Anesth Analg. 2017 Feb;124(2):524-530. doi: 10.1213/ANE.0000000000001424. PMID 27537927
- [Background] Silva YR, Li SK, Rickard MJ. Does the addition of deep breathing exercises to physiotherapy-directed early mobilisation alter patient outcomes following high-risk open upper abdominal surgery? Cluster randomised controlled trial. Physiotherapy. 2013 Sep;99(3):187-93. doi: 10.1016/j.physio.2012.09.006. Epub 2012 Dec 1. PMID 23206316
- [Background] Souza Possa S, Braga Amador C, Meira Costa A, Takahama Sakamoto E, Seiko Kondo C, Maida Vasconcellos AL, Moran de Brito CM, Pereira Yamaguti W. Implementation of a guideline for physical therapy in the postoperative period of upper abdominal surgery reduces the incidence of atelectasis and length of hospital stay. Rev Port Pneumol. 2014 Mar-Apr;20(2):69-77. doi: 10.1016/j.rppneu.2013.07.005. Epub 2013 Nov 27. PMID 24290563
- [Background] Browning L, Denehy L, Scholes RL. The quantity of early upright mobilisation performed following upper abdominal surgery is low: an observational study. Aust J Physiother. 2007;53(1):47-52. doi: 10.1016/s0004-9514(07)70061-2. PMID 17326738